CLINICAL TRIAL: NCT01168921
Title: A Phase II Trial of Eltrombopag for Patients With Chronic Lymphocytic Leukemia (CLL) and Thrombocytopenia
Brief Title: Phase II Eltrombopag in Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0123; NCI-2012-01905 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-02

CONDITIONS: CLL; Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; Thrombocytopenia; Small lymphocytic lymphoma; SLL; Eltrombopag; Promacta; thrombopoietin (TPO)-receptor agonist; platelets
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Thrombocytopenia; Jacobs syndrome | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eltrombopag (Experimental): Starting dose 75 mg by mouth (PO) daily for 28 day cycle.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Starting dose 75 mg by mouth (PO) daily for 28 day cycle
  Other Names: Promacta

SUMMARY:
The goal of this clinical research study is to learn if eltrombopag can help to increase the number of platelets in patients with CLL. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

When the number of platelets in your body gets too low, it can cause bleeding, which may cause serious health problems and/or prevent you from receiving chemotherapy. Eltrombopag is designed to act like a protein in your body that helps make platelets. This may help increase your platelet counts.

Study Drug Administration:

You will take pills of the study drug by mouth 1 time each day on an empty stomach (1 hour before or 2 hours after a meal). You should take the pills with 1 cup (8 ounces) of water. You should wait at least 4 hours between taking eltrombopag and eating foods with calcium (dairy products and/or juices with added calcium) or taking drugs/supplements with iron, calcium, aluminum, magnesium, selenium and/or zinc. Other drugs may also affect eltrombopag. Be sure to tell your doctor about any drugs and/or supplements you may be taking.

During your study visits, your doctor will check your platelet counts to see if they improve. If they do not improve, your dose of study drug may be increased. Your doctor will instruct you on each dose of eltrombopag you should take.

Do not take more than 1 dose of eltrombopag on any one day. If you forget to take a dose, you should skip the missed dose and continue your regular dosing schedule. Do not take a double dose to make up for a missed one.

Study Visits:

Each study "cycle" will be 28 days.

Each week during Cycle 1, then every 2 weeks during Cycles 2 and 3:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any bleeding that may have occurred since the last study visit.
* Blood (about 1 tablespoon) will be drawn for routine tests.

On Day 1 (+/- 7 days) of Cycles 4 and beyond:

* You will have a physical exam.
* You will be asked about any bleeding that may have occurred since the last study visit.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will also have a bone marrow aspirate/biopsy to check the status of the disease and to check your platelet counts. This test will only be performed every 3 cycles.

Length of Study Participation:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if you require other treatment for CLL or if intolerable side effects occur.

Follow-Up:

After you stop taking eltrombopag for any reason, your platelet counts may drop. This may increase your risk of bleeding. Blood (about 1 tablespoon) will be drawn each week for 4 weeks to check your platelet counts.

This is an investigational study. Eltrombopag is FDA approved and commercially available for use in chronic immune thrombocytopenic purpura (ITP - severe bleeding due to platelet destruction by the immune system). The use of this drug in patients with CLL is investigational.

Up to 36 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL)
2. Age >/= 18 years
3. PLT transfusion-dependent, defined as need for transfusion to maintain PLT count >/=20K/µL, or the average of two (non-transfused) PLT counts taken within 2 weeks of the screening period </=50K/µL, with no individual count >55K/µL
4. Patients with ITP must have failed at least 1 prior treatment for ITP including one of the following: corticosteroids, rituximab, splenectomy, cyclosporine
5. At least 3 weeks must have elapsed since the last chemotherapy treatment for CLL
6. ECOG performance status (PS) </=2
7. Adequate liver function (total bilirubin </=2* upper limit normal (ULN); ALT </=2.5* ULN)
8. Adequate renal function (serum creatinine Cr </=2.2 mg/dL)
9. For patients with ITP on corticosteroids or cyclosporine, dose of corticosteroids or cyclosporine must be stable for 2 weeks prior to enrollment and planned to be tapered in patients responding to eltrombopag
10. Able to provide informed consent

Exclusion Criteria:

1. Concurrent chemotherapy for CLL
2. Diagnosis of Richter's transformation
3. Uncontrolled autoimmune hemolytic anemia i.e. patients with AIHA that is not controlled with treatment such as corticosteroids or cyclosporine. This would include patients who require PBRC transfusions or who do not have a stable hemoglobin (HGB) due to ongoing hemolysis.
4. Concurrent treatment for ITP (except for corticosteroids and cyclosporine)
5. Diagnosis of myelodysplastic syndrome or acute myeloid leukemia
6. Active infection or significant medical illness as determined by the treating physician
7. Treatment with thrombomimetic agents in the past 3 months (rTPO, PEG-rHuMGDF, Nplate or Promacta)
8. Pregnant or breast feeding subjects and subjects not willing to use adequate contraceptive precautions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-11-03 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G. Wierda, MD, PHD, BS, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eltrombopag
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eltrombopag
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 62 [47 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: Response is Complete Response (CR) + Major Response (MR). Complete response was defined as an increase in platelet count to ≥100K/µL for at least 4 weeks. Major response was defined as an increase in platelet count from <20K/µL to ≥20K/μL and by at least 100% for at least 8 weeks; or for pts starting with >20K/μL platelet count, absolute increase in platelet count of ≥30K/μL for at least 4 weeks.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 23
Participants | 12

2. Secondary Outcome: Time to CLL Progression Requiring Leukemia Treatment
Description: The number of months from start of treatment to CLL progression, requiring leukemia treatment. Disease Progression (PD) is defined as a >/= 50% increase in at least one of the following in responding participants: >/= 2 lymph nodes (on 2 exams 2 weeks apart), liver or spleen (below costal margin) , or absolute number of circulating lymphocytes (>/= 10L/ul).
Time Frame: Up to 4 years
Measure: Median (Full Range); unit: Months
Arm/Group | Eltrombopag
Number analyzed (Participants) | 23
Months | 5.8 [2.8 to 21]

ADVERSE EVENTS:
Time Frame: Up to 4 years
Arm/Group | Eltrombopag
All-Cause Mortality (participants affected / at risk) | 2/23
Serious Adverse Events (participants affected / at risk) | 6/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eltrombopag (N=23)
Weakness (General disorders) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)
Flu (General disorders) | 1 (1)
Altered Mental Status (Psychiatric disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (4)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Splenectomy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eltrombopag (N=23)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 23 (52)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Bronchitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-12-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT01168921/Prot_SAP_000.pdf